CLINICAL TRIAL: NCT03394118
Title: A Phase II Study for Evaluating Anti-tumor Efficacy of TAGRISSO (Osimertinib) in NSCLC Patients in Whom T790 Mutations Are Detected by Liquid Biopsy Using Bronchoalveolar Lavage Fluid, Plasma or Pleural Effusion
Brief Title: TAGRISSO (Osimertinib) in NSCLC Patients in Whom T790 Mutations Are Detected by Liquid Biopsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Chang-Min Choi, Associate professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2016-00578_ESR-16-11898
Record Dates: First submitted 2017-08-01; First posted 2018-01-09 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: NSCLC
Keywords: T790 mutation; Liquid biopsy
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group_TAGRISSO (Experimental): Each subject will continue the study drug(Osimertinib) until disease progression or manifestation of unacceptable toxicity during the study period.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — A cycle of study treatment is defined as 28 days. Each subject will continue the study drug(Osimertinib) until disease progression or manifestation of unacceptable toxicity during the study period. The study drug will be administered orally as one 80 mg tablet once a day. The initial dose of the study drug 80 mg daily can be reduced to 40 mg once daily.

SUMMARY:
In this trial, anti-tumor efficacy of TAGRISSO in NSCLC patients in whom T790 mutations are detected by liquid biopsy.

DETAILED DESCRIPTION:
This study is designed to be a phase II, Open-label, single-arm, single-center study to evaluate anti-tumor efficacy of TAGRISSO in NSCLC patients in whom T790 mutations are detected by liquid biopsy using at least one of the samples such as plasma, bronchoalveolar lavage fluid, and pleural effusion. Approximately 63 patients will be enrolled into the trial, and expected study duration is 43 months from IRB and Korea: MFDA approval date.

Each subject will continue the study drug (Osimertinib) until disease progression or manifestation of unacceptable toxicity during the study period. The study drug will be administered orally as one 80 mg tablet once a day. The initial dose of the study drug 80 mg daily can be reduced to 40 mg once daily.

A cycle of study treatment is defined as 28 days. Patients will be enrolled for 31 months and will be followed-up regularly, and duration of follow-up for each patient will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20, and patients who understand information about the trial and voluntarily agree to participate in the trial
2. Histological or cytological confirmation diagnosis of NSCLC and inoperable stage IIIB or IV at the time of study enrolment
3. Patients with EGFR sensitizing mutation (E19Del, L858R, L861Q, G719X) positive, who had shown clinical benefits (responders (CR or PR) and SD ≥6 months) from EGFR-TKIs and had developed progressive disease following those therapy

   * Patients who have histories of previous exposure to EGFR-TKIs or other systemic chemotherapies are permitted (regardless of the order of treatment)
   * Treated with at least one of KGFR-TKIs (regardless of treatment with or without systemic chemotherapies)
   * In case the patient previously received any of the treatments including systemic chemotherapy, radiation therapy, surgery, and hormonal therapy, there should be at least 2 weeks of time interval between the last day of the previous treatment and the start of TAGRISSO™, and the remaining toxicity should be ≤ CTCAE grade 1 at the time of starting study treatment (except alopecia and grade 2, prior platinum-therapy related neuropathy)
4. ECOG performance status 0-2
5. Patients in whom T790 mutations are detected in at least one of the samples including tumor tissues, BALF (cell-free DNA), plasma (cell-free DNA), and pleural effusion (cell-free DNA)
6. At least one measurable lesions according to RECIST v 1.1
7. Female with childbearing potential (within 1 year of time interval between last menses and the date of informed consent) who use appropriate contraception methods and are not on breast-feeding, and tested negative for pregnancy test or are sure to have a proof for infertility prior to drug initiation
8. Males willing to use barrier contraception methods during study period (Patients should inform their sexual partners of the use of the allowed contraception methods.)
9. Patients willing to provide informed consent with date and signature included prior to all study-specific procedures, samplings and analyse
10. Patients who have proper organ functions as follows:

    * ANC ≥ 1500/mm3,
    * PLT counts ≥ 100,000/mm3,
    * Hb ≥ 9.0g/dL,
    * Serum creatinine ≤ upper normal limit,
    * AST/ ALT/ ALP ≤ 3 times upper normal limit, Total bilirubin ≤2.0mg/dL (In case of liver metastasis AST/ ALT/ ALP ≤ 5 times upper normal limit, in case of bone metastasis, ALP ≤ 5 times upper normal limit)
11. Patients must have a life expectancy ≥ 12 weeks

Exclusion Criteria:

1. Patients who were previously treated with any of the drugs targeting T790M mutation such as AZD9291 (Osimertinib), HM61713 (Olmutinib), and CO-1686 (Rociletinib)
2. Patients currently receiving medications known to be potent inhibitors of CYP3A4 and potent inducers of CYP3A4 (at least 1week prior study enrolment)
3. Patients who have preexisting or coexisting malignancies in other parts except for effectively treated non-melanoma skin cancer, CIS cervical cancer, DCIS breast cancer, thyroid cancer or malignancies that were effectively treated, have maintained at least 3 years of remission state and can be regarded as completely cured
4. Patients who have severe or unstable medical conditions such as prior or current clinically significant cardiovascular abnormality in accordance with the investigator's judgment such as uncontrolled hypertension, heart failure (NYHA classification ≥3), unstable angina or uncontrolled arrhythmia, and acute myocardial infarction within 6 months before study enrolment corrected QTcB >450msec in 12 lead EKG
5. Patients with current or prior interstitial lung disease
6. Patients with current or prior uncontrolled gastrointestinal diseases (e.g., crohn's disease, ulcerative colitis, chronic diarrhea, malabsorption) that would preclude adequate absorption of IP.
7. Patients with active hepatitis B (identified by the presence of HBsAg and/or HBV DNA), active hepatitis C (identified by the presence of HCV RNA), and known human immunodeficiency virus (HIV)
8. Patients with histories of hypersensitivity to IP or any components of the agent
9. Patients with any of the following genetic predispositions including galactose intolerance, lactose intolerance, or glucose-galactose malabsorption
10. Patients with symptomatic CNS metastases who are neurologically unstable (Cases with radiologically and neurologically stable disease after discontinuation of the administration of corticosteroids and anticonvulsants for at least 4 weeks are excluded)
11. Patients with uncontrolled infective diseases (Patients who require non-oral antibiotics injection must be excluded, but they can be included if the diseases are completely resolved.)
12. Patients who are difficult or unlikely to comply with study procedures, restrictions, requirements, and follow-up managements according to the investigator's judgment
13. Patients who were administered other study drugs within 30 days before starting the study treatment (Patients are permitted if they were given any of the drugs including gefitinib, erlotinib, and afatinib)
14. Patients with any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia and grade 2, prior platinum-therapy related neuropathy.
15. Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
ORR | through study completion (43 months)
  Objective response rate (ORR) including rate of CR and PR on based of RECIST 1.1

SECONDARY OUTCOMES:
DCR | through study completion (43 months)
  Disease control rate (DCR) including rate of CR, PR and SD on based of RECIST 1.1
PFS | through study completion (43 months)
  Progression-free survival (PFS) the time from first dose of the study drug until the date of disease progression or death by any cause.
T790M postive rate in Plasma cell free DNA | through study completion (43 months)
T790M postive rate in BALF free DNA | through study completion (43 months)
T790M postive rate in tissue | through study completion (43 months)
Concordance rate of T790M positivity between plasma & BALF | through study completion (43 months)
T790M sensitivity & specificity in Plasma & BALF (gold standard: tissue biopsy) | through study completion (43 months)
The frequency of occurrence of grade 3 or higher AE/SAEs | through study completion (43 months)
  AE/SAE assessement on the base of NCI-CTCAE (version 4.03).

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Min Cho, Ph. D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided